CLINICAL TRIAL: NCT01853748
Title: A Randomized Phase II Study of Trastuzumab Emtansine (T-DM1) vs. Paclitaxel in Combination With Trastuzumab for Stage I HER2-Positive Breast Cancer (ATEMPT Trial)
Brief Title: T-DM1 vs Paclitaxel/Trastuzumab for Breast (ATEMPT Trial)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Sara Tolaney, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-048
Record Dates: First submitted 2013-04-24; First posted 2013-05-15 (Estimated); Results first posted 2022-01-19 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Paclitaxel; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trastuzumab emtansine (T-DM1) (Active Comparator): T-DM1 3.6mg/kg every three weeks by IV for 17 doses for a total of 51 weeks
  Interventions: Drug: Trastuzumab emtansine
- Paclitaxel + Trastuzumab (Active Comparator): paclitaxel 80 mg/m2 IV weekly and trastuzumab 4 mg/kg IV load, followed by 2 mg/kg IV weekly for 12 weeks, followed by trastuzumab 6 mg/kg IV every 3 weeks for 13 treatments
  Interventions: Drug: Trastuzumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Trastuzumab
  Arms: Paclitaxel + Trastuzumab
Drug: Paclitaxel
  Arms: Paclitaxel + Trastuzumab
Drug: Trastuzumab emtansine
  Other Names: T-DM1
  Arms: Trastuzumab emtansine (T-DM1)

SUMMARY:
This research study is a Phase II clinical trial. Phase II clinical trials test the effectiveness of an investigational drug to learn whether the drug works in treating a specific cancer. "Investigational" means that the drug is still being studied and that research doctors are trying to find out more about it-such as the safest dose to use, the side effects it may cause, and if the drug is effective for treating different types of cancer. It also means that the FDA has not approved this drug for use patients undergoing adjuvant treatment for HER2+ breast cancer. Trastuzumab emtansine (T-DM1) is a drug that may stop cancer cells from growing. This drug has been used in other research studies and information from those other research studies suggests that this drug may help to prevent the recurrence of breast cancer in this research study.

The use of T-DM1 in this research study is experimental, which means it is not approved by any regulatory authority for the adjuvant treatment of HER2-positive breast cancer. However, it FDA-approved for metastatic HER2-positive breast cancer. T-DM1 has caused cancer cells to die in laboratory studies. In preclinical studies, this drug has prevented or slowed the growth of breast cancer. The breast cancer treatments (paclitaxel and Trastuzumab) used in this study are considered part of standard-of-care regimens in early breast cancer. A standard treatment means that this is a treatment that would be accepted by the majority of the medical community as a suitable treatment for your type of breast cancer.

In this research study, the investigators are looking to see if the study drug T-DM1 will have less side effects than traditional HER2-positive breast cancer treatment of trastuzumab and paclitaxel. The investigators are also hoping to learn about the long term benefits and disease-free survival of participants who take the study drug T-DM1 in comparison to those participants to take the combination of trastuzumab and paclitaxel.

DETAILED DESCRIPTION:
If a participant agrees to participate in this study she will be asked to undergo some screening tests or procedures to confirm that she is eligible. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if turns out that she does not take part in this research study. If she has had some of these tests or procedures recently, they may or may not have to be repeated. These tests and procedures will include: a medical history, performance status, assessment of your tumor, blood tests, cardiac tests, pregnancy test and a collection of tumor tissue. If these tests show that she is eligible to participate in the research study, she will begin the study treatment. If she does not meet the eligibility criteria, she will not be able to participate in this research study.

Because no one knows which of the study options is best, the participant will be "randomized" into one of the study groups after she has had her breast surgery: Group 1 or Group 2. Randomization means that she is put into a group by chance. Neither the participant nor the research doctor will choose what group she will be in. The participant will have a one in three chance of being placed in any group. Approximately 375 study participants will receive the study drug, while 125 study participants will receive the standard therapy of trastuzumab and paclitaxel.

Group 1 participants will receive the study drug T-DM1 every three weeks by IV (intravenous injection) for 17 treatments (total of 51 weeks).

Group 2 participants will receive the FDA-approved drugs Paclitaxel and Trastuzumab once per week by IV for 12 weeks. Then beginning week 13, participants will receive Trastuzumab only by IV injection every three weeks for the next 13 treatments.

During all cycles the participant will have a physical exam and tumor assessment.

The investigators would like to keep track of the participant's medical condition for the next five years after the final dose of study drug. The investigators would like to do this by regular visits every 6 months for 3 years after completion of study treatment, and then once a year for the next two years. The investigators may ask for additional follow-up by phone after completion of these visits.

Participants who undergo lumpectomy (breast conserving surgery) need to receive breast radiation therapy to participate in this study. Participants who have undergone a mastectomy may receive chest wall and lymph node radiation (as determined by discussion with their physician). Radiation Therapy will begin after the conclusion of all study paclitaxel doses, and after 12 weeks fo the study drug T-DM1.

ELIGIBILITY:
Inclusion Criteria:

* HER2-positive Stage I histologically confirmed invasive carcinoma of the breast
* ER/PR determination is required
* HER2 positive, confirmed by central testing: IHC 3+, FISH HER2/CEP17 <2.0 with an average HER2 copy number >/=6.0, or FISH HER2/CEP17 >/= 2.0
* Bilateral breast cancers that individually meet eligibility criteria are allowed
* Subjects with multifocal or multicentric disease are eligible as long as each tumor individually meets eligibility criteria
* Subjects with a history of ipsilateral DCIS are eligible if they were treated with wide-excision alone, without radiation therapy; Patients with a history of contralateral DCIS are not eligible.
* Should have tumor tissue available and a tissue block of sufficient size to make 15 slides, which must be sent to a DFCI site for testing
* Less than or equal to 90 days since most recent breast surgery for this breast cancer
* All tumor should be removed by either a modified radical mastectomy or a segmental mastectomy (lumpectomy) with either a sentinel node biopsy or axillary dissection
* All margins should be clear of invasive cancer or DCIS
* May have received up to 4 weeks of tamoxifen therapy or other hormonal therapy, for adjuvant therapy for this cancer
* Prior oophorectomy for cancer prevention is allowed
* Subjects who have undergone partial breast radiation (duration </= 7 days) prior to registration are eligible. Partial breast radiation must be completed prior to 2 weeks before starting protocol therapy.
* Must have discontinued any investigational drug at least 2 weeks prior to participation
* Willing to use one highly effective from of nonhormonal contraception or two effective forms of nonhormonal contraception while on study and for 7 months after end of study treatment
* Subjects undergoing lumpectomy must have no contraindications to radiation therapy

Exclusion Criteria:

* Pregnant or breastfeeding
* Use of potent CYP3A4 inhibitors during the study treatment period
* Excessive alcohol intake (more than 3 alcoholic beverages per day)
* Locally advanced tumors at diagnosis
* History of previous invasive breast cancer
* History of prior chemotherapy in the past 5 years
* History of prior trastuzumab or prior paclitaxel therapy
* Active, unresolved infection
* Active liver disease
* History of a different malignancy except for the following: disease free for at least 5 years and at low risk for recurrence; cervical cancer in situ, basal or squamous cell carcinoma of the skin
* Active cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2013-05; Primary Completion 2019-08-26 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tolaney, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (85):
- United States (85):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - Hartford Hospital, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - Hartford Healthcare Cancer Institute at The Hospital of Central Connecticut, New Britain, Connecticut
  - William W Backus Hospital, Norwich, Connecticut
  - Georgetown Hospital, Washington D.C., District of Columbia
  - Washington Cancer Institute at Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Mountain States Tumor Institute, Boise, Idaho
  - Mountain States Tumor Institute, Fruitland, Idaho
  - Mountain States Tumor Institute, Meridian, Idaho
  - Mountain States Tumor Institute, Nampa, Idaho
  - Mountain States Tumor Institute, Twin Falls, Idaho
  - Loyola University Medical Center, Maywood, Illinois
  - University of Chicago Comprehensive Cancer Center at Silver Cross Hospital, New Lenox, Illinois
  - University of Chicago Medical Center for Advanced Care Orland Park, Orland Park, Illinois
  - Indiana University - Wishard Hospital, Indianapolis, Indiana
  - Indiana University Health - Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Indiana University Health - University Hospital, Indianapolis, Indiana
  - Indiana University - Springmill Medical Clinic, Indianapolis, Indiana
  - Eastern Maine Medical Center's Cancer Care, Brewer, Maine
  - Johns Hopkins - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Suburban Hospital Cancer Program, Bethesda, Maryland
  - Johns Hopkins - Green Spring Station, Lutherville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute at Faulkner Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mass General North Shore Cancer Center, Danvers, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Dana-Farber Cancer Institute at Milford Hospital, Milford, Massachusetts
  - Univeristy of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Siteman Cancer Center - St. Peters, City of Saint Peters, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University, School of Medicine, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Siteman Cancer Center - West County, St Louis, Missouri
  - New Hampshire Oncology-Hematology, PA, Concord, New Hampshire
  - New Hampshire Oncology-Hematology, PA, Hooksett, New Hampshire
  - New Hampshire Oncology-Hematology, PA, Laconia, New Hampshire
  - Dana-Farber Cancer Insitute at Londonderry Hospital, Londonderry, New Hampshire
  - Memorial Sloan Kettering Cancer Center-Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center-Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center Westchester, Harrison, New York
  - Queens Hospital Center, Comprehensive Cancer Center, Jamaica, New York
  - Northwell Health/Monter Cancer Center, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center-Mercy, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center-Sleepy Hollow, Sleepy Hollow, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Rex Cancer Center, Raleigh, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Lehigh Valley Hospital/Lehigh Valley Health Network, Allentown, Pennsylvania
  - UPMC/HVHS Cancer Center, UPMC Beaver, Beaver, Pennsylvania
  - UPMC CancerCenters Butler, Butler, Pennsylvania
  - UPMC Horizon (Shenango), Farrell, Pennsylvania
  - Arnold Palmer Cancer Center-Greensburg, Greensburg, Pennsylvania
  - Arnold Palmer Medical Oncology Oakbrook, Greensburg, Pennsylvania
  - UPMC Horizon (Greenville), Greenville, Pennsylvania
  - UPMC Pinnacle Harrisburg, Harrisburg, Pennsylvania
  - UPMC Cancer Center Jefferson Regional Med Ctr, Jefferson Hills, Pennsylvania
  - UPMC Conemaugh Cancer Center, Johnstown, Pennsylvania
  - UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC East, Monroeville, Pennsylvania
  - Arnold Palmer Medical Oncology-Mt Pleasant, Mount Pleasant, Pennsylvania
  - UPMC Jameson Cancer Center, New Castle, Pennsylvania
  - UPMC St. Margaret, Pittsburgh, Pennsylvania
  - UPMC Cancer Center St. Clair Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Shadyside, Pittsburgh, Pennsylvania
  - UPMC Passavant, Pittsburgh, Pennsylvania
  - UPMC Northwest (Franklin), Seneca, Pennsylvania
  - UPMC Northwest (Oil City), Seneca, Pennsylvania
  - UPMC and the Washington Hospital Center, Washington, Pennsylvania
  - Tennessee Oncology/Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Baylor College of Medicine-Baylor Clinic, Houston, Texas
  - Harris County Hospital District-Ben Taub General Hospital, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Harris County Hospital District-Smith Clinic, Houston, Texas
  - University of Washington Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- [Derived] Tarantino P, Tayob N, Villacampa G, Dang C, Yardley DA, Isakoff SJ, Valero V, Faggen M, Mulvey T, Bose R, Weckstein D, Wolff AC, Reeder-Hayes K, Rugo HS, Ramaswamy B, Zuckerman D, Hart L, Gadi VK, Constantine M, Cheng K, Garrett AM, Marcom PK, Albain K, DeFusco P, Tung N, Ardman B, Nanda R, Jankowitz RC, Rimawi M, Abramson V, Pohlmann PR, Van Poznak C, Forero-Torres A, Liu MC, Ruddy KJ, Waks AG, DeMeo M, Burstein HJ, Partridge AH, Dell'Orto P, Russo L, Krause E, Newhouse DJ, Kurt BB, Mittendorf EA, Schneider B, Prat A, Winer EP, Krop IE, Tolaney SM; Consortium of the TBCRC Translational Investigators; TBCRC Translational Investigators. Adjuvant Trastuzumab Emtansine Versus Paclitaxel Plus Trastuzumab for Stage I Human Epidermal Growth Factor Receptor 2-Positive Breast Cancer: 5-Year Results and Correlative Analyses From ATEMPT. J Clin Oncol. 2024 Nov;42(31):3652-3665. doi: 10.1200/JCO.23.02170. Epub 2024 Jun 27. PMID 38935923
- [Derived] Sella T, Zheng Y, Tayob N, Ruddy KJ, Freedman RA, Dang C, Yardley D, Isakoff SJ, Valero V, DeMeo M, Burstein HJ, Winer EP, Wolff AC, Krop I, Partridge AH, Tolaney SM. Treatment discontinuation, patient-reported toxicities and quality-of-life by age following trastuzumab emtansine or paclitaxel/trastuzumab (ATEMPT). NPJ Breast Cancer. 2022 Nov 30;8(1):127. doi: 10.1038/s41523-022-00495-x. PMID 36450763
- [Derived] Barroso-Sousa R, Tarantino P, Tayob N, Dang C, Yardley DA, Isakoff SJ, Valero V, Faggen M, Mulvey T, Bose R, Hu J, Weckstein D, Wolff AC, Reeder-Hayes K, Rugo HS, Ramaswamy B, Zuckerman D, Hart L, Gadi VK, Constantine M, Cheng K, Briccetti F, Schneider B, Garrett AM, Marcom K, Albain K, DeFusco P, Tung N, Ardman B, Nanda R, Jankowitz RC, Rimawi M, Abramson V, Pohlmann PR, Van Poznak C, Forero-Torres A, Liu M, Ruddy KJ, Zheng Y, Rosenberg SM, Gelber RD, Trippa L, Barry W, DeMeo M, Burstein H, Partridge A, Winer EP, Krop I, Tolaney SM. Cardiac outcomes of subjects on adjuvant trastuzumab emtansine vs paclitaxel in combination with trastuzumab for stage I HER2-positive breast cancer (ATEMPT) study (TBCRC033): a randomized controlled trial. NPJ Breast Cancer. 2022 Feb 16;8(1):18. doi: 10.1038/s41523-022-00385-2. PMID 35173164
- [Derived] Tolaney SM, Tayob N, Dang C, Yardley DA, Isakoff SJ, Valero V, Faggen M, Mulvey T, Bose R, Hu J, Weckstein D, Wolff AC, Reeder-Hayes K, Rugo HS, Ramaswamy B, Zuckerman D, Hart L, Gadi VK, Constantine M, Cheng K, Briccetti F, Schneider B, Garrett AM, Marcom K, Albain K, DeFusco P, Tung N, Ardman B, Nanda R, Jankowitz RC, Rimawi M, Abramson V, Pohlmann PR, Van Poznak C, Forero-Torres A, Liu M, Ruddy K, Zheng Y, Rosenberg SM, Gelber RD, Trippa L, Barry W, DeMeo M, Burstein H, Partridge A, Winer EP, Krop I. Adjuvant Trastuzumab Emtansine Versus Paclitaxel in Combination With Trastuzumab for Stage I HER2-Positive Breast Cancer (ATEMPT): A Randomized Clinical Trial. J Clin Oncol. 2021 Jul 20;39(21):2375-2385. doi: 10.1200/JCO.20.03398. Epub 2021 Jun 2. PMID 34077270

RESULTS

PARTICIPANT FLOW:
Groups:
- Paclitaxel + Trastuzumab (TH): paclitaxel 80 mg/m2 IV weekly and trastuzumab 4 mg/kg IV load, followed by 2 mg/kg IV weekly for 12 weeks, followed by trastuzumab 6 mg/kg IV every 3 weeks for 13 treatments
Period: Allocation
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab (TH)
Started | 384 | 128
Completed | 383 | 114
Not Completed | 1 | 14
Not completed — Withdrawal by Subject | 1 | 13
Not completed — not sufficient to receive intervention | 0 | 1
Period: Follow-Up
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab (TH)
Started | 383 | 114
Completed | 293 | 97
Not Completed | 90 | 17
Not completed — Withdrawal by Subject | 7 | 6
Not completed — Adverse Event | 67 | 7
Not completed — not available for data collection | 16 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab (TH) | Total
Number analyzed (Participants) | 383 | 114 | 497
Age, Continuous [Median (Full Range); unit: Years] | 56 [32 to 85] | 55 [23 to 82] | 56 [23 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 383 | 114 | 497
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 327 | 93 | 420
  Black or African American | 21 | 7 | 28
  Asian | 22 | 4 | 26
  More than one race | 2 | 1 | 3
  Other | 11 | 9 | 20
Region of Enrollment [Number; unit: participants]
  United States | 383 | 114 | 497

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants of Clinically Relevant Toxicities (CRT)
Description: Clinically relevant toxicities will include the composite incidence of grade 3 or higher non-hematologic toxicity, grade 2 or higher neurotoxicity, and grade 4 or higher hematologic toxicity. These toxicities will only be assessed at the pre-specified toxicity-assessment visits. In addition, the following events, regardless of timing of their occurrence, will also count towards the composite endpoint: febrile neutropenia, any toxicity requiring dose-delay, discontinuation of any study treatment (Paclitaxel, Trastuzumab, or T-DM1) for toxicity, and any serious adverse event (SAE).
Time Frame: 5 years after completion of study treatment or until death, whichever occurs first.
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab
Number analyzed (Participants) | 383 | 114
Participants
  Grade 3 or higher non-hematologic toxicity | 36 | 13
  Grade 2 or higher neurotoxicity | 42 | 26
  Grade 4 or higher hematologic toxicity | 4 | 0
  Febrile neutropenia | 0 | 2
  Any toxicity requiring dose delay | 106 | 30
  Any toxicity requiring early discontinuation of protocol therapy | 67 | 7
  Serious adverse event | 11 | 6

2. Primary Outcome: 3-year Disease Free Survival (DFS) Rate of Trastuzumab Emtansine (TDM-1)
Description: Disease-free survival (DFS) is evaluated and defined per protocol: from the time of randomization until the to the occurrence of the first of the following events:
  * Local/regional recurrence: a recurrent or new invasive ipsilateral breast cancer, invasive breast cancer in the axilla, regional lymph nodes, chest wall, or skin of the ipsilateral breast.
  * Contralateral invasive breast cancer,
  * Distant recurrence: metastatic disease that has either been biopsy confirmed or clinically diagnosed as recurrent invasive breast cancer. A single new lesion on a bone scan without evidence of lytic disease on x-ray and without symptoms does not in and of itself constitute distant recurrence, but multiple new bone lesions, or increased isotope uptake associated with new bone symptoms are more likely due to metastases. Bone metastases must be documented with x-rays and clinical description.
  * Death from any cause
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab
Number analyzed (Participants) | 383 | 114
proportion of participants | 0.978 [0.963 to 0.993] | 0.934 [0.889 to 0.988]

3. Secondary Outcome: Incidence Rate of Grade 3-4 Treatment-Related Toxicity
Description: All grade 3 - 4 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv4 as reported on case report forms were counted. Incidence is the number of patients experiencing at least one treatment-related grade >=3 AE of any type during the time of observation.
Time Frame: AE is reported every 3 weeks for the first 12 weeks, then every 9 weeks for the subsequent 39 weeks, then follow-up up to 5 years after completion of study treatment or until death, whichever occurs first. Median follow-up 3.1 years.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab
Number analyzed (Participants) | 383 | 114
proportion of participants | 0.16 [0.12 to 0.2] | 0.23 [0.15 to 0.32]

4. Secondary Outcome: Quality of Life (QOL) FACT B Total Score at Baseline
Description: The QOL assessments questionnaire should be completed via the tablet provided by the study or on any available computer with an internet connection. The FACT-B questionnaire consists of five subscale, listed below:
  Physical well being(PWB): range 0-28 Social/Family well being(SWB): range 0-28 Emotional well being(EWB): range 0-24 Functional well being(FWB): range 0-28 Breast cancer subscale(BCS): range 0-40 The total score (FACTB) is calculated by summarizing all the subscales listed above, therefore it ranges from 0 to 148. The higher the score the better the outcome (applies to all sub-scales as well).
Time Frame: at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab (TH)
Number analyzed (Participants) | 351 | 103
score on a scale | 126.25 (14.29) | 116.69 (19.03)

5. Secondary Outcome: Quality of Life (QOL) FACT B Total Score at Week 3
Description: as for outcome 4
Time Frame: at week 3
Population: not all patients required to complete the QOL
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab
Number analyzed (Participants) | 326 | 89
score on a scale | 127.07 (14.52) | 116.6 (18.9)

6. Secondary Outcome: Quality of Life (QOL) FACT B Total Score at Week 12
Description: as for outcome 4
Time Frame: at week 12
Population: not all patients required to complete the QOL
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab
Number analyzed (Participants) | 302 | 83
score on a scale | 124.36 (16.3) | 108.25 (23.33)

7. Secondary Outcome: Quality of Life (QOL) FACT B Total Score at 6 Months
Description: as for outcome 4
Time Frame: at 6 months
Population: not all patients required to complete the QOL
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab
Number analyzed (Participants) | 299 | 83
score on a scale | 123 (16.71) | 118.16 (21.73)

8. Secondary Outcome: Quality of Life (QOL) FACT B Total Score at 1 Year
Description: as for outcome 4
Time Frame: at 1 year
Population: not all patients required to complete the QOL
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab
Number analyzed (Participants) | 276 | 87
score on a scale | 123.29 (16.44) | 120.3 (20.88)

9. Secondary Outcome: Quality of Life (QOL) FACT B Total Score at 18 Months
Description: as for outcome 4
Time Frame: at 18 months
Population: not all patients required to complete the QOL
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab
Number analyzed (Participants) | 279 | 77
score on a scale | 126.42 (15.67) | 117.93 (23.55)

10. Secondary Outcome: Quality of Life (QOL) FACT B Total Score at 24 Months
Description: as for outcome 4
Time Frame: at 24 months
Population: not all patients required to complete the QOL
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab
Number analyzed (Participants) | 260 | 71
score on a scale | 127.19 (16.16) | 121.73 (22.00)

11. Secondary Outcome: Number of Patients Has Neuropathy
Description: Neuropathy evaluated by Patient Neurotoxicity Questionnaire (PNQ) defined per protocol.
Time Frame: Surveys are took at week 3, 12 and month 6 and 12 during treatment, and month 18. The data cutoff date is 18 month.
Population: The PNQ analysis was done on patients that completed at least baseline questionnaires and at least one follow-up questionnaire. Some patients did not complete this questionnaire at either baseline or follow-up. This is the reason for the reduced number of patients when reporting PNQ results.
Measure: Count of Participants; unit: Participants
Groups:
- T-DM1 With no Baseline Neuropathy: T-DM1 3.6mg/kg every three weeks by IV for 17 doses for a total of 51 weeks. No neuropathy at baseline
- TH With no Baseline Neuropathy: paclitaxel 80 mg/m2 IV weekly and trastuzumab 4 mg/kg IV load, followed by 2 mg/kg IV weekly for 12 weeks, followed by trastuzumab 6 mg/kg IV every 3 weeks for 13 treatments.
  No neuropathy at baseline
- T-DM1 With Any Baseline Neuropathy: T-DM1 3.6mg/kg every three weeks by IV for 17 doses for a total of 51 weeks. Neuropathy at baseline
- TH With Any Baseline Neuropathy: paclitaxel 80 mg/m2 IV weekly and trastuzumab 4 mg/kg IV load, followed by 2 mg/kg IV weekly for 12 weeks, followed by trastuzumab 6 mg/kg IV every 3 weeks for 13 treatments.
  Neuropathy at baseline
Arm/Group | T-DM1 With no Baseline Neuropathy | TH With no Baseline Neuropathy | T-DM1 With Any Baseline Neuropathy | TH With Any Baseline Neuropathy
Number analyzed (Participants) | 291 | 81 | 58 | 23
Participants
  No, mild, or moderate neuropathy | 267 | 64 | 36 | 11
  Moderate to severe and severe neuropathy | 24 | 17 | 22 | 12
Statistical Analysis 1: Comparison: T-DM1 With no Baseline Neuropathy vs TH With no Baseline Neuropathy vs T-DM1 With Any Baseline Neuropathy vs TH With Any Baseline Neuropathy; Test type: Superiority; p = 0.0012, Mantel Haenszel

12. Secondary Outcome: Percentage of Work Time Missed Because of Health
Description: Effects of therapy on work productivity and activity - work time missed because of health, evaluated using the Work Productivity and Activity Impairment Questionnaire (WPAI-SHP), which defined per protocol.
Time Frame: Surveys are took at week 3, 12 and month 6 and 12 during treatment, and month 18, 24, 30 and 36 during follow up.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab
Number analyzed (Participants) | 383 | 114
percentage of time
  Baseline | 22 (35) | 25 (34)
  3 weeks | 13 (28) | 27 (36)
  12 weeks | 9 (21) | 22 (33)
  6 months | 8 (21) | 7 (18)
  12 months | 8 (21) | 8 (20)
  18 months | 3 (13) | 4 (16)

13. Secondary Outcome: Percentage of Impairment While Working Because of Health (Mean, SD)
Description: Effects of therapy on work productivity and activity - Impairment While Working because of health, evaluated using the Work Productivity and Activity Impairment Questionnaire (WPAI-SHP), which defined per protocol.
Time Frame: Surveys are took at week 3, 12 and month 6 and 12 during treatment, and month 18, 24, 30 and 36 during follow up.
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- Trastuzumab Emtansine (T-DM1): T-DM1 3.6mg/kg every three weeks by IV for 17 doses for a total of 51 weeks
  Trastuzumab emtansine
- Paclitaxel + Trastuzumab: paclitaxel 80 mg/m2 IV weekly and trastuzumab 4 mg/kg IV load, followed by 2 mg/kg IV weekly for 12 weeks, followed by trastuzumab 6 mg/kg IV every 3 weeks for 13 treatments
  Trastuzumab
  Paclitaxel
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab
Number analyzed (Participants) | 383 | 114
percentage of time
  Baseline | 10 (18) | 20 (26)
  3 weeks | 9 (16) | 21 (25)
  12 weeks | 11 (18) | 21 (26)
  6 months | 9 (14) | 11 (19)
  12 months | 12 (20) | 9 (18)
  18 months | 3 (8) | 8 (17)

14. Secondary Outcome: Percentage of Overall Work Impairment Because of Health
Description: Effects of therapy on work productivity and activity - Work Impairment because of health, evaluated using the Work Productivity and Activity Impairment Questionnaire (WPAI-SHP), which defined per protocol.
Time Frame: Surveys are took at week 3, 12 and month 6 and 12 during treatment, and month 18, 24, 30 and 36 during follow up.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab (TH)
Number analyzed (Participants) | 383 | 114
percentage of time
  Baseline | 19 (26) | 31 (31)
  3 weeks | 14 (23) | 30 (29)
  12 weeks | 16 (22) | 29 (29)
  6 months | 13 (18) | 14 (22)
  12 months | 16 (24) | 13 (22)
  18 months | 4 (12) | 9 (18)

15. Secondary Outcome: Percentage of Activity Impairment Because of Health
Description: Effects of therapy on work productivity and activity - Activity Impairment because of health, evaluated using the Work Productivity and Activity Impairment Questionnaire (WPAI-SHP), which defined per protocol.
Time Frame: Surveys are took at week 3, 12 and month 6 and 12 during treatment, and month 18, 24, 30 and 36 during follow up.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab (TH)
Number analyzed (Participants) | 383 | 114
percentage of time
  Baseline | 14 (22) | 22 (26)
  3 weeks | 12 (19) | 22 (27)
  12 weeks | 13 (19) | 33 (31)
  6 months | 15 (21) | 17 (22)
  12 months | 15 (21) | 14 (23)
  18 months | 7 (17) | 15 (27)

16. Secondary Outcome: Number of Patients Have Alopecia
Description: alopecia assessment is a 5-item questionnaire that will assess the impact alopecia has had on these patients and will be conducted electronically at pre-specified study visits. If electronic evaluation is not possible, paper evaluation will be conducted.
Time Frame: Median follow-up was 3.9 years. The AE data cutoff date is 21 April 2020.
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab
Number analyzed (Participants) | 383 | 114
Participants | 157 | 0
Statistical Analysis 1: Comparison: Trastuzumab Emtansine (T-DM1) vs Paclitaxel + Trastuzumab; Test type: Superiority; p = 0.0001, Regression, Linear

17. Secondary Outcome: 3-year T-DM1 iDFS Percentage by Tumor Size and Hormone Receptor (HR) Status
Description: Disease-free survival (DFS) is evaluated in patients treated with trastuzumab emtansine, which is defined per protocol: from the time of randomization until the to the occurrence of the first of the following events:
  * Local/regional recurrence: a recurrent or new invasive ipsilateral breast cancer, invasive breast cancer in the axilla, regional lymph nodes, chest wall, or skin of the ipsilateral breast.
  * Contralateral invasive breast cancer,
  * Distant recurrence: metastatic disease that has either been biopsy confirmed or clinically diagnosed as recurrent invasive breast cancer. A single new lesion on a bone scan without evidence of lytic disease on x-ray and without symptoms does not in and of itself constitute distant recurrence, but multiple new bone lesions, or increased isotope uptake associated with new bone symptoms are more likely due to metastases. Bone metastases must be documented with x-rays and clinical description.
  * Death from any cause
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Trastuzumab Emtansine (T-DM1) With Tumor Size < 1 cm; Trastuzumab Emtansine (T-DM1) With Tumor Size >= 1 cm: T-DM1 3.6mg/kg every three weeks by IV for 17 doses for a total of 51 weeks
Arm/Group | Trastuzumab Emtansine (T-DM1) With Tumor Size < 1 cm | Trastuzumab Emtansine (T-DM1) With Tumor Size >= 1 cm
Number analyzed (Participants) | 163 | 220
percentage of participants | 98.7 [96.9 to 100] | 97.2 [95 to 99.4]

18. Secondary Outcome: Number of Incidence of Grade 3-4 Cardiac Left Ventricular Dysfunction
Description: as for outcome 3
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab (TH)
Number analyzed (Participants) | 383 | 114
Participants | 3 | 2

19. Secondary Outcome: Number of Incidence of T-DM1 Induced Grade 2-3 Thrombocytopenia
Description: Reversible Grade 1-4 thrombocytopenia has been observed in ongoing studies with trastuzumab emtansine.
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab
Number analyzed (Participants) | 383 | 114
Participants | 42 | 1
Statistical Analysis 1: Comparison: Trastuzumab Emtansine (T-DM1) vs Paclitaxel + Trastuzumab; Test type: Superiority; p = 0.0001, Fisher Exact

20. Secondary Outcome: Number of SNPs With Top Associations of Trastuzumab Emtansine-induced Grade 2-4 Thrombocytopenia in the T-DM1 Arm
Description: DNA will be genotyped for SNPs and CNV markers using the Infinium Human Omni1 array (1.2 million SNP platform) from Illumina. A gene-based association analyses for thrombocytopenia or bleeding is applied with significancy (p-value). This analysis was only conducted in the T-DM1 arm.
Time Frame: DNA sample collected at pre-treatment. AE is reported every 3 weeks for the first 12 weeks, then every 9 weeks for the subsequent 39 weeks.
Measure: Number; unit: number of SNPs
Arm/Group | Trastuzumab Emtansine (T-DM1)
Number analyzed (Participants) | 110
number of SNPs | 54

21. Secondary Outcome: Percentage of Patients With Amenorrhea
Description: All grade 3 - 4 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv4 as reported on case report forms were counted. Incidence is the number of patients experiencing at least one treatment-related grade >=3 AE of any type during the time of observation.
  For those who were premenopausal pre-chemotherapy, at each follow-up visit (every six months) in order to assess for duration of amenorrhea and also premature ovarian failure.
Time Frame: Surveys are took at month 6 and 12 during treatment, and month 18, 24, 30 and 36 during follow up.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab (TH)
Number analyzed (Participants) | 383 | 114
percentage of participants
  6 months | 80 | 21
  1 year | 71 | 22
  18 months | 64 | 20
  24 months | 74 | 15
  30 months | 60 | 11
  36 months | 45 | 9

22. Secondary Outcome: Gene Mutation Assessed Using High-throughput Mutation Profiling System (Oncomap)
Description: Archival tumor tissue from all patients will be assessed using a high-throughput mutation profiling system (Oncomap) to query a large panel of cancer gene mutations.
Time Frame: After treatment
Population: no genomic data were collected using the Oncomap system
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab (TH)
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Median Overall Survival (OS)
Description: OS is evaluated in patients with Stage I HER2-positive breast cancer treated with trastuzumab emtansine
Time Frame: Reported every 3 weeks for the first 12 weeks, then every 9 weeks for the subsequent 39 weeks, then follow-up up to 5 years after completion of study treatment or until death, whichever occurs first.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab (TH)
Number analyzed (Participants) | 383 | 114
months | NA [NA to NA] — The cohorts have good overall survival outcome, and never reached the median survival. The overall survival rate at month 80, the longest follow up time of the cohort, is 98%. Therefore, the median survival and the corresponding 95% CI can not be estimated. | NA [NA to NA] — The cohorts have good overall survival outcome, and never reached the median survival. The overall survival rate at month 80, the longest follow up time of the cohort, is 98%. Therefore, the median survival and the corresponding 95% CI can not be estimated.

ADVERSE EVENTS:
Time Frame: AE is reported every 3 weeks for the first 12 weeks, then every 9 weeks for the subsequent 39 weeks, then follow-up up to 5 years after completion of study treatment or until death, whichever occurs first. Median follow-up 3.1 years. The AE data cutoff date is 21 April 2020.
Arm/Group | Trastuzumab Emtansine (T-DM1) | Paclitaxel + Trastuzumab
All-Cause Mortality (participants affected / at risk) | 6/383 | 1/114
Serious Adverse Events (participants affected / at risk) | 62/383 | 26/114
Other Adverse Events (participants affected / at risk) | 383/383 | 114/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Emtansine (T-DM1) (N=383) | Paclitaxel + Trastuzumab (N=114)
Anemia (Blood and lymphatic system disorders) | 4 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0
Fatigue (General disorders) | 3 | 2
Infusion related reaction (General disorders) | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Oral hemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Gum infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1
CPK increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 3 | 7
Platelet count decreased (Investigations) | 12 | 0
Weight loss (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 9 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Irregular menstruation (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Premature menopause (Reproductive system and breast disorders) | 1 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0
Hot flashes (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 8 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Emtansine (T-DM1) (N=383) | Paclitaxel + Trastuzumab (N=114)
Ear pain (Ear and labyrinth disorders) | 4 | 0
Hearing impaired (Ear and labyrinth disorders) | 6 | 0
Tinnitus (Ear and labyrinth disorders) | 3 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 4 | 1
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 53 | 26
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 2 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 4 | 0
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 9 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 1 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 14 | 3
Pericardial effusion (Cardiac disorders) | 1 | 1
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 3
Sinus tachycardia (Cardiac disorders) | 3 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Cardiac disorders - Other (Cardiac disorders) | 3 | 1
Chills (General disorders) | 29 | 3
Edema face (General disorders) | 4 | 3
Edema limbs (General disorders) | 35 | 19
Edema trunk (General disorders) | 1 | 1
Facial pain (General disorders) | 3 | 0
Fatigue (General disorders) | 250 | 80
Fever (General disorders) | 39 | 9
Flu like symptoms (General disorders) | 24 | 5
Gait disturbance (General disorders) | 0 | 2
Infusion related reaction (General disorders) | 23 | 11
Injection site reaction (General disorders) | 1 | 0
Irritability (General disorders) | 3 | 2
Localized edema (General disorders) | 11 | 4
Non-cardiac chest pain (General disorders) | 12 | 2
Pain (General disorders) | 46 | 23
General disorders and administration site conditions - Other (General disorders) | 17 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 21 | 64
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 29 | 15
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 4 | 0
Erythroderma (Skin and subcutaneous tissue disorders) | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 2
Hypohidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 4 | 14
Nail loss (Skin and subcutaneous tissue disorders) | 4 | 5
Nail ridging (Skin and subcutaneous tissue disorders) | 6 | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 2 | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 10
Rash acneiform (Skin and subcutaneous tissue disorders) | 30 | 16
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 39 | 17
Scalp pain (Skin and subcutaneous tissue disorders) | 1 | 4
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 10 | 3
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 3 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 53 | 20
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0
Endocrine disorders - Other (Endocrine disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 30 | 7
Bloating (Gastrointestinal disorders) | 7 | 4
Cecal hemorrhage (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 1
Colonic ulcer (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 111 | 12
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 63 | 54
Dry mouth (Gastrointestinal disorders) | 118 | 6
Duodenal hemorrhage (Gastrointestinal disorders) | 2 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 47 | 15
Dysphagia (Gastrointestinal disorders) | 2 | 1
Esophagitis (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 6 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 47 | 18
Gastrointestinal pain (Gastrointestinal disorders) | 4 | 2
Gingival pain (Gastrointestinal disorders) | 3 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 6 | 2
Mucositis oral (Gastrointestinal disorders) | 48 | 15
Nausea (Gastrointestinal disorders) | 192 | 46
Oral dysesthesia (Gastrointestinal disorders) | 0 | 2
Oral hemorrhage (Gastrointestinal disorders) | 7 | 0
Oral pain (Gastrointestinal disorders) | 2 | 3
Periodontal disease (Gastrointestinal disorders) | 3 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 8 | 2
Stomach pain (Gastrointestinal disorders) | 4 | 1
Tooth development disorder (Gastrointestinal disorders) | 1 | 0
Tooth discoloration (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 38 | 13
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 19 | 5
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 7 | 1
Allergic reaction (Immune system disorders) | 9 | 1
Cytokine release syndrome (Immune system disorders) | 1 | 0
Immune system disorders - Other (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bladder infection (Infections and infestations) | 1 | 0
Breast infection (Infections and infestations) | 5 | 2
Bronchial infection (Infections and infestations) | 2 | 1
Catheter related infection (Infections and infestations) | 1 | 1
Conjunctivitis infective (Infections and infestations) | 2 | 0
Esophageal infection (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 1 | 2
Gum infection (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 2 | 0
Lip infection (Infections and infestations) | 1 | 0
Lip infection (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 5 | 1
Mucosal infection (Infections and infestations) | 2 | 1
Nail infection (Infections and infestations) | 2 | 1
Otitis externa (Infections and infestations) | 3 | 0
Otitis media (Infections and infestations) | 7 | 1
Papulopustular rash (Infections and infestations) | 7 | 5
Paronychia (Infections and infestations) | 3 | 0
Pharyngitis (Infections and infestations) | 2 | 1
Phlebitis infective (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 1 | 0
Rhinitis infective (Infections and infestations) | 4 | 0
Rhinitis infective (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 15 | 1
Sinusitis (Infections and infestations) | 15 | 3
Skin infection (Infections and infestations) | 4 | 2
Skin infection (Infections and infestations) | 12 | 7
Soft tissue infection (Infections and infestations) | 1 | 0
Stoma site infection (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 4 | 2
Upper respiratory infection (Infections and infestations) | 13 | 2
Upper respiratory infection (Infections and infestations) | 28 | 9
Urinary tract infection (Infections and infestations) | 2 | 3
Urinary tract infection (Infections and infestations) | 34 | 3
Vaginal infection (Immune system disorders) | 1 | 1
Vaginal infection (Infections and infestations) | 6 | 2
Wound infection (Infections and infestations) | 2 | 0
Infections and infestations - Other (Infections and infestations) | 13 | 10
Ankle fracture (Infections and infestations) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 15 | 0
Burn (Injury, poisoning and procedural complications) | 5 | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 44 | 13
Fall (Injury, poisoning and procedural complications) | 5 | 5
Fracture (Injury, poisoning and procedural complications) | 1 | 3
Intraoperative breast injury (Injury, poisoning and procedural complications) | 0 | 1
Intraoperative skin injury (Injury, poisoning and procedural complications) | 0 | 1
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 3 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 5 | 1
Alanine aminotransferase increased (Investigations) | 111 | 18
Alkaline phosphatase increased (Investigations) | 57 | 2
Aspartate aminotransferase increased (Investigations) | 129 | 9
Blood bilirubin increased (Investigations) | 38 | 4
Creatinine increased (Investigations) | 4 | 5
Ejection fraction decreased (Investigations) | 3 | 2
Lipase increased (Investigations) | 2 | 0
Lymphocyte count decreased (Investigations) | 14 | 4
Lymphocyte count increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 24 | 18
Platelet count decreased (Investigations) | 89 | 5
Weight gain (Investigations) | 8 | 6
Weight loss (Investigations) | 28 | 6
White blood cell decreased (Investigations) | 24 | 14
Investigations - Other, specify (Investigations) | 9 | 3
Anorexia (Metabolism and nutrition disorders) | 58 | 14
Dehydration (Metabolism and nutrition disorders) | 10 | 4
Glucose intolerance (Metabolism and nutrition disorders) | 3 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 9 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 28 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 5 | 1
Hypernatremia (Metabolism and nutrition disorders) | 3 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 19 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 5
Hypoglycemia (Metabolism and nutrition disorders) | 9 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 4
Hypokalemia (Metabolism and nutrition disorders) | 32 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 11 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 94 | 28
Arthritis (Musculoskeletal and connective tissue disorders) | 7 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 12
Bone pain (Musculoskeletal and connective tissue disorders) | 13 | 6
Chest wall pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 9 | 6
Growth suppression (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 8 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 75 | 15
Neck pain (Musculoskeletal and connective tissue disorders) | 11 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 6 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 34 | 14
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 29 | 5
Akathisia (Nervous system disorders) | 2 | 2
Amnesia (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 4 | 1
Concentration impairment (Nervous system disorders) | 4 | 1
Dizziness (Nervous system disorders) | 28 | 15
Dysgeusia (Nervous system disorders) | 55 | 11
Dysphasia (Nervous system disorders) | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 118 | 33
Hypersomnia (Nervous system disorders) | 2 | 0
Lethargy (Nervous system disorders) | 1 | 0
Leukoencephalopathy (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 8 | 4
Paresthesia (Nervous system disorders) | 28 | 7
Peripheral motor neuropathy (Nervous system disorders) | 23 | 17
Peripheral sensory neuropathy (Nervous system disorders) | 119 | 50
Presyncope (Nervous system disorders) | 3 | 1
Sinus pain (Nervous system disorders) | 1 | 1
Spasticity (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 2 | 1
Nervous system disorders - Other (Nervous system disorders) | 7 | 6
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Blurred vision (Eye disorders) | 25 | 6
Cataract (Eye disorders) | 2 | 0
Conjunctivitis (Eye disorders) | 1 | 2
Dry eye (Eye disorders) | 44 | 5
Eye pain (Eye disorders) | 2 | 1
Floaters (Eye disorders) | 2 | 0
Retinal detachment (Eye disorders) | 1 | 0
Retinal tear (Eye disorders) | 1 | 0
Retinal vascular disorder (Eye disorders) | 0 | 1
Watering eyes (Eye disorders) | 12 | 3
Eye disorders - Other (Eye disorders) | 16 | 5
Agitation (Psychiatric disorders) | 4 | 0
Anxiety (Psychiatric disorders) | 38 | 23
Confusion (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 34 | 8
Hallucinations (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 58 | 30
Libido decreased (Psychiatric disorders) | 3 | 2
Restlessness (Psychiatric disorders) | 2 | 0
Psychiatric disorders - Other (Psychiatric disorders) | 3 | 4
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 21 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 56 | 21
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 27 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 90 | 25
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 45 | 10
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 15 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 21 | 8
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 17 | 6
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 5 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal calculi (Renal and urinary disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 7 | 2
Urinary incontinence (Renal and urinary disorders) | 3 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 8 | 0
Urinary urgency (Renal and urinary disorders) | 3 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 2 | 0
Breast pain (Reproductive system and breast disorders) | 31 | 7
Dysmenorrhea (Reproductive system and breast disorders) | 1 | 0
Dyspareunia (Reproductive system and breast disorders) | 2 | 0
Genital edema (Reproductive system and breast disorders) | 0 | 1
Irregular menstruation (Reproductive system and breast disorders) | 13 | 2
Menorrhagia (Reproductive system and breast disorders) | 9 | 1
Ovarian rupture (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 0
Uterine hemorrhage (Reproductive system and breast disorders) | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 4 | 0
Vaginal dryness (Reproductive system and breast disorders) | 18 | 8
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 | 0
Vaginal pain (Reproductive system and breast disorders) | 1 | 1
Vaginal stricture (Reproductive system and breast disorders) | 0 | 1
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 14 | 2
Flushing (Vascular disorders) | 4 | 6
Hematoma (Vascular disorders) | 3 | 0
Hot flashes (Vascular disorders) | 60 | 34
Hypertension (Vascular disorders) | 78 | 29
Hypotension (Vascular disorders) | 2 | 1
Lymphedema (Vascular disorders) | 8 | 5
Phlebitis (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT01853748/Prot_SAP_000.pdf